CLINICAL TRIAL: NCT00159250
Title: Restoring Dystrophin Expression in Duchenne Muscular Dystrophy: A Phase I/II Clinical Trial Using AVI-4658
Brief Title: Safety and Efficacy Study of Antisense Oligonucleotides in Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Department of Health, United Kingdom (Other Government); Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 05/MRE12/32; AVI-4658-33 (Other: Sarepta); 2006-003833-33 (EudraCT Number)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy;; antisense oligonucleotides;; gene restoration;; deletion
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — eteplirsen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose (Experimental): Low dose of AVI-4658
  Interventions: Drug: AVI-4658 (PMO)
- High dose (Experimental): High dose of AVI-4658
  Interventions: Drug: AVI-4658 (PMO)

INTERVENTIONS:
Drug: AVI-4658 (PMO) — morpholino antisense oligonucleotide

SUMMARY:
Duchenne muscular dystrophy (DMD), a fatal muscle degenerative disorder, arises from mutations in the dystrophin gene. Antisense therapy with the use of antisense oligonucleotides (AON) has the potential to restore effectively the production of dystrophin, the defective protein, in >70% of DMD. This could result in increased life expectancy through improved muscle survival and function. Recent scientific research has demonstrated the potential of this technique to skip mutated dystrophin exons, restore the reading frame and generate functional dystrophin protein. Having demonstrated proof-of-principle in human cell culture and animal model studies, we now intend to determine efficacy and safety of this approach to induce dystrophin exon skipping in children with DMD.

The specific aim of this phase I/II study is to assess efficacy (dystrophin production) and safety of intramuscular administered morpholino oligomer directed against exon 51 (AVI-4658 PMO). We are performing parallel preclinical studies to develop methods of systemic delivery that will be necessary for future phase II/III clinical studies.

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is the most common form of muscular dystrophy affecting 1 in every 3500 live male births. The disease is characterised by severe muscle wasting and weakness, which becomes clinically evident between the ages of 3 to 5 years. Affected individuals stop walking by 12 years of age and usually do not survive beyond the age of 20 unless ventilated. In general DMD is caused by mutations that disrupt the reading frame thus leading to a failure to express dystrophin.

Recent scientific research has led to the belief that DMD may be treated by correcting the genetic error in the dystrophin gene which causes DMD. Most children with DMD have a deletion, i.e., a mutation which removes part of the dystrophin gene. A novel technique using antisense technology to skip a specific exon and bypass faulty genetic material, thus allowing production of functional dystrophin to be produced, has been developed.These antisense oligonucleotides (AON) target and bypass faulty genetic material and allow production of functional protein.This has been successfully demonstrated in cultured human DMD cells and in mouse and canine DMD models.The restored production of dystrophin is predicted to reduce muscle pathology significantly.

In the early part of the study we compared different antisense oligomers chemical modification and concluded that the morpholino backbone is significantly superior when administered to skeletal muscle compared to a number of other types of antisense.

The aim of this phase I/II clinical study is to assess efficacy and safety of AVI-4658, a morpholino antisense directed against exon 51, in DMD individuals with deletions which would benefit from skipping exon 51.

The proposed work is presented in 4 sections detailing the main approaches.

Study design

This dose escalation IM trial will involve of up to 9 subjects, subdivided in three groups, of three subjects each. Patients in group 1 will be recruited sequentially whilst patients in groups 2 and 3 will be recruited serially.

* Group 1 (3 patients) will receive intramuscular administration of a low concentration of study drug (extensor digitorum brevis muscle, EDB) and will undergo a muscle biopsy between days 14 and 28 after intramuscular (IM) administration of the AVI-4658.
* Group 2 (3 patients) will undergo an identical procedure but receiving an intermediate dose of the AVI-4658.
* Group 3 (3 patients) will be recruited to receive the highest dose of the AVI-4658 but only if the results in the first 2 cohort of patients show a lack of efficacy of the lower doses. Up to an additional 3 subjects may be enrolled in cohorts 1 or 2, should cohort 3 not be enrolled.

Screening

* A physical examination, including body weight, height, arm span, neuromuscular examination and vital signs (blood pressure, pulse, respiration, and temperature).
* Neuropsychiatric assessment of both subject and the family.
* Molecular genetic on blood sample and dystrophin analysis of original muscle biopsy obtained at diagnosis.
* Muscle MRI scans of lower limbs to assess the preservation of the muscle to be targeted with the injection of AON.
* Biochemical (blood) and urine investigation to include standard biochemistry and haematology (full blood count; coagulation screen; liver function test; serum Ig; protein electrophoresis; inflammatory markers; creatinine kinase; gamma glutamyl transferase; urine biochemistry).
* Cardiovascular assessments: ECG and heart echocardiogram.
* Pulmonary assessments: Forced vital capacity, overnight oxygen saturation monitoring.
* Skin biopsy for MyoD-transfection.

Procedure

* The muscle to be used is the extensor digitorum brevis, a foot muscle with very little function in children with mobility difficulties.
* Local injection will be performed directly through the skin using a combined EMG-delivery needle. While the procedure could be performed under local anaesthetic; where possible, it will be performed under general anaesthetic in order to reduce distress to the subject. A skin tattoo featuring a 1 cm x 1 cm grid with 2 lines in between to divide it in 9 smaller squares will be used to mark the site of the injection precisely and for a subsequent muscle biopsy.
* The total volume of each injection will be 100 μL containing the AVI-4658. Nine injections will be performed at 3 mm intervals inside the 1 cm2 grid tattoo. The depth of the injection will be carefully recorded.

Observation

* Patients will be closely monitored within the clinical research facility by designated nursing staff educated in the trial protocol and with experience in similar Phase I/II studies.
* The clinical research facility has close access to intensive care unit facilities in the event of an unforeseen adverse reaction.

Follow-up Day 2 - Patients will be discharged. Prior to discharge, a brief physical examination and systems review will be performed.

Day 3 - A further brief physical examination and systems review including examination of the injection sites and reporting of any reactions. This examination can be performed at the local surgery or at the hospital of the referring clinician.

Days 5, 7 - Contact with the subject and inquire as to current status.

Day 14 to 28 - The subject is admitted to hospital. Perform systems assessment (physical examination), body weight and vital signs. Blood and urine biochemistry will be repeated then as well as open biopsies of both injected muscles will be performed under general or local anaesthetic.

Day 30 - Contact with the subject and inquiry as to current status.

Day 60 - Contact the subject and inquiry as to current status.

Day 120 - (Final Visit at the hospital where the study drug was administered). A brief physical examination and systems review will be performed.

MDEX Consortium.

The PRECLINICAL studies were performed by the following groups, who are all members of the MDEX consortium:

1. Prof Francesco Muntoni, Dr. Jennifer Morgan. Dubowitz Neuromuscular Centre, Department of Paediatrics, Imperial College Hammersmith Hospital Campus, Du Cane Road London W12 ONN
2. Prof Dominic Wells; Dr Kim Wells. Gene Targeting Group, Department of Cellular and Molecular Neuroscience Division of Neuroscience and Mental Health, Imperial College, Charing Cross Campus, St. Dunstan's Road, London W6 8RP
3. Prof George Dickson; Dr Ian Graham. Gene Therapy Laboratory, Centre for Biomedical Sciences, Royal Holloway - University of London, Egham
4. Dr Matthew Wood. Department of Physiology, Anatomy and Genetics, South Parks Road,Oxford OX1 3QX, United Kingdom (UK).
5. Professor Steve Wilton. Experimental Molecular Medicine Group, Centre for Neuromuscular and Neurological Disorders, University of Western Australia

Additional CLINICAL SUPPORT other than the Study officials will be provided by:

Dubowitz Neuromuscular Centre, Department of Paediatrics, Hammersmith Hospital Campus, Du Cane Road, W12ONN: Prof Caroline Sewry; Dr. Maria Kinali; Dr Virginia Arechavala; Dr Lucy Feng

Department of Surgery, St Mary's Hospital Trust, Imperial College Praed Street, London, W2 1NY: Mr David Hunt

DNA Laboratory, Genetics Centre, 5th Floor Guy's Tower, Guy's Hospital London SE1 9RT: Dr Steve Abbs

Academic Unit of Child and Adolescent Psychiatry, Division of Neuroscience and Mental Health, Imperial College, St Mary's Campus, Norfolk Place, Paddington,London, W2 1PG: Professor Elena Garralda

MDEX Study coordinator:

Dr K Ganeshaguru, Dubowitz Neuromuscular Centre, Department of Paediatrics, Hammersmith Hospital Campus, Imperial College London, Du Cane Road, W12ONN, k.ganeshaguru@imperial.ac.uk

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male ≥ 10 years and ≤ 17 years of age at the time of study drug administration.
2. Subject has clinical diagnosis compatible with Duchenne's Muscular Dystrophy (DMD) and evidence of mutational and dystrophin defects from muscle biopsy consistent with DMD (out-of frame deletions, absent dystrophin).Eligible deletions are those that can be rescued by the skipping of exon 51 [45-50; 47-50; 48-50; 49-50; 50; 52; 52-63].
3. Subject has had a muscle biopsy analysed, showing <5% revertant fibres present. Biopsy may be collected at the time of DMD diagnosis or as part of protocol screening procedures.
4. Subject is unable to ambulate or stand independently.
5. Subject has Stage 1 to 3 EDB muscle preservation determined by MRI.
6. Subject has a forced vital capacity ≥ 25% confirmed within 3 months from Day One.
7. Subject has mean oxygen saturation monitoring > 94% in overnight domiciliary overnight sleep study within 3 months of Day One.
8. Subject has the ability to comply with all study evaluations and return for all study.
9. Subject and parent have psychiatric adjustments, adequately supportive psychosocial circumstances and a full understanding of study aims process and likely outcomes.

Exclusion Criteria:

1. Subject has had external digitorum brevis (EDB) muscle removed.
2. Subject has Stage 4 EDB muscle preservation determined by MRI.
3. Subject has a left ventricular shortening fraction of < 25% and/or an ejection fraction of < 35% by echocardiography at visit one or within three months of visit one.
4. Subject has evidence of nocturnal hypoventilation (mean oxygen saturation at night of ≤ 94%) confirmed via overnight sleep study at Visit One (as screening procedure) or within 3 months of Visit One by overnight sleep study.
5. Subject has severe respiratory insufficiency defined by the need for invasive or non-invasive mechanical ventilation (does not include nocturnal ventilatory support).
6. Subject has severe cognitive dysfunction rendering them unable to understand and collaborate with study protocol.
7. Subject has immune deficiency or autoimmune disease.
8. Subject has a known bleeding disorder or has received chronic anticoagulant treatment within three months of study entry.
9. Subject has received pharmacologic treatment, apart from corticosteroids, that might affect muscle strength or function within 8 weeks of study entry (viz.,anabolic steroids, creatine protein supplementation, albuterol or other beta agonists).
10. Subject has had surgery within 3 months of study entry or planned for anytime during study.
11. Subject has active significant illness at time of study entry.
12. Subject has is unable to undergo MRI testing (viz., has metal implants).
13. Subject or parent has active psychiatric disorder, has adverse psychosocial circumstances, recent significant emotional loss, history of depressive or anxiety disorders that might interfere with protocol completion or compliance.
14. Subject has any known allergies to products likely to be used in the study (viz.,antiseptics, anaesthetics).
15. Subject has used any experimental treatments or has participated in any clinical trial within 4 weeks of study entry.
16. Subject has used intranasal, inhaled or topical steroids for a condition other than muscular dystrophy within 1 weeks of study entry.

Ages: 10 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — male
Enrollment: 7 (Actual)
Dates: Start 2007-10-26 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2009-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Muntoni, FRCPCH, Principal Investigator — Dubowitz neuromuscular Centre, Imperial College, London; Kate Bushby, MRCP, Study Director — Institute of Human Genetics, University of Newcastle upon Tyne; Volker Straub, FRCPCH, Study Director — Institute of Human Genetics, University of Newcastle upon Tyne
Locations (1):
- Dubowitz Neuromuscular Centre, Hammersmith Hospital and Clinical Trails Unit, St Mary's Hospital, London, United Kingdom

REFERENCES:
- [Background] Lu QL, Morris GE, Wilton SD, Ly T, Artem'yeva OV, Strong P, Partridge TA. Massive idiosyncratic exon skipping corrects the nonsense mutation in dystrophic mouse muscle and produces functional revertant fibers by clonal expansion. J Cell Biol. 2000 Mar 6;148(5):985-96. doi: 10.1083/jcb.148.5.985. PMID 10704448
- [Background] De Angelis FG, Sthandier O, Berarducci B, Toso S, Galluzzi G, Ricci E, Cossu G, Bozzoni I. Chimeric snRNA molecules carrying antisense sequences against the splice junctions of exon 51 of the dystrophin pre-mRNA induce exon skipping and restoration of a dystrophin synthesis in Delta 48-50 DMD cells. Proc Natl Acad Sci U S A. 2002 Jul 9;99(14):9456-61. doi: 10.1073/pnas.142302299. Epub 2002 Jun 20. PMID 12077324
- [Background] Lu QL, Mann CJ, Lou F, Bou-Gharios G, Morris GE, Xue SA, Fletcher S, Partridge TA, Wilton SD. Functional amounts of dystrophin produced by skipping the mutated exon in the mdx dystrophic mouse. Nat Med. 2003 Aug;9(8):1009-14. doi: 10.1038/nm897. Epub 2003 Jul 6. PMID 12847521
- [Background] Lu QL, Rabinowitz A, Chen YC, Yokota T, Yin H, Alter J, Jadoon A, Bou-Gharios G, Partridge T. Systemic delivery of antisense oligoribonucleotide restores dystrophin expression in body-wide skeletal muscles. Proc Natl Acad Sci U S A. 2005 Jan 4;102(1):198-203. doi: 10.1073/pnas.0406700102. Epub 2004 Dec 17. PMID 15608067
- [Background] Gebski BL, Mann CJ, Fletcher S, Wilton SD. Morpholino antisense oligonucleotide induced dystrophin exon 23 skipping in mdx mouse muscle. Hum Mol Genet. 2003 Aug 1;12(15):1801-11. doi: 10.1093/hmg/ddg196. PMID 12874101
- [Background] Fletcher S, Honeyman K, Fall AM, Harding PL, Johnsen RD, Wilton SD. Dystrophin expression in the mdx mouse after localised and systemic administration of a morpholino antisense oligonucleotide. J Gene Med. 2006 Feb;8(2):207-16. doi: 10.1002/jgm.838. PMID 16285002
- [Background] Alter J, Lou F, Rabinowitz A, Yin H, Rosenfeld J, Wilton SD, Partridge TA, Lu QL. Systemic delivery of morpholino oligonucleotide restores dystrophin expression bodywide and improves dystrophic pathology. Nat Med. 2006 Feb;12(2):175-7. doi: 10.1038/nm1345. Epub 2006 Jan 29. PMID 16444267
- [Result] Kinali M, Arechavala-Gomeza V, Feng L, Cirak S, Hunt D, Adkin C, Guglieri M, Ashton E, Abbs S, Nihoyannopoulos P, Garralda ME, Rutherford M, McCulley C, Popplewell L, Graham IR, Dickson G, Wood MJ, Wells DJ, Wilton SD, Kole R, Straub V, Bushby K, Sewry C, Morgan JE, Muntoni F. Local restoration of dystrophin expression with the morpholino oligomer AVI-4658 in Duchenne muscular dystrophy: a single-blind, placebo-controlled, dose-escalation, proof-of-concept study. Lancet Neurol. 2009 Oct;8(10):918-28. doi: 10.1016/S1474-4422(09)70211-X. Epub 2009 Aug 25. PMID 19713152

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose AVI-4658: Low dose of AVI-4658
  0.09 mg doses were diluted in 900 μL normal saline (0·9%) and injected to the extensor digitorum brevis (EDB) muscle
- High Dose AVI-4658: High dose of AVI-4658
  0.9 mg doses were diluted in 900 μL normal saline (0·9%) and injected to the extensor digitorum brevis (EDB) muscle
Period: Overall Study
Arm/Group | Low Dose AVI-4658 | High Dose AVI-4658
Started | 2 | 5
Completed | 2 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose AVI-4658 | High Dose AVI-4658 | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 5 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 14.5 [13 to 16] | 11.8 [10 to 15] | 13.1 [10 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 5 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 | 5 | 7
Mobility [Count of Participants; unit: Participants]
  Wheelchair for 11 years | 1 | 0 | 1
  Wheelchair for 10 years; rides static bike for 10 | 1 | 0 | 1
  Wheelchair for 10 years | 0 | 1 | 1
  Walks indoors | 0 | 1 | 1
  Walks unaided | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Related to AVI-4568
Description: Number of Subjects with Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Time Frame: Baseline up to Day 120
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose AVI-4658 | High Dose AVI-4658
Number analyzed (Participants) | 2 | 5
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Injection Site Reactions
Time Frame: From the Day of Screening to Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose AVI-4658 | High Dose AVI-4658
Number analyzed (Participants) | 2 | 5
Participants | 2 | 4

3. Primary Outcome: Number of Subjects With Clinically Significant Change From Baseline in Laboratory Values
Description: Assessed by light microscopy and immunocytochemistry to detect the differences in inflammatory infiltrates between the AVI-4568 and placebo-treated EDB muscles
Time Frame: From the Day of Screening up to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose AVI-4658 | High Dose AVI-4658
Number analyzed (Participants) | 2 | 5
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Induced Skipping of Exon 51 in the Treated Extensor Digitorum Brevis (EDB) Muscle Determined by Reverse Transcription Polymerase Chain Reaction
Description: Induced Skipping of Exon 51 in the Treated Extensor Digitorum Brevis (EDB) Muscle Determined by Reverse Transcription Polymerase Chain Reaction was assessed by Sequencing of the RT-PCR products
Time Frame: Day 14 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose AVI-4658 | High Dose AVI-4658
Number analyzed (Participants) | 2 | 5
Participants | 2 | 5

5. Secondary Outcome: Number of Participants With Restoration of Dystrophin Protein Expression Measured by Immunocytochemistry
Time Frame: Day 14 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose AVI-4658 | High Dose AVI-4658
Number analyzed (Participants) | 2 | 5
Participants | 0 | 5

6. Secondary Outcome: Number of Participants With Restoration of Dystrophin Protein Expression Measured by Western Blot Analysis
Time Frame: Day 14 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose AVI-4658 | High Dose AVI-4658
Number analyzed (Participants) | 2 | 5
Participants | 0 | 5

ADVERSE EVENTS:
Time Frame: 120 days
Arm/Group | Low Dose AVI-4658 | High Dose AVI-4658
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 2/2 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose AVI-4658 (N=2) | High Dose AVI-4658 (N=5)
Bilateral erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
Myoglobinuria (Immune system disorders) | 0 (0) | 3 (3)
Bilateral oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decline in cardiac function (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes